CLINICAL TRIAL: NCT03010696
Title: The Correlation Between Gut Microbiome/Metabolite and End Stage Renal Disease (ESRD)
Status: Completed | Type: Observational
Sponsor: China Agricultural University (Other)
Collaborators: Peking University Aerospace Center Hospital (Other); General Hospital of Chinese Armed Police Forces (Other); Beijing Anzhen Hospital (Other); Peking University Shougang Hospital (Other); Beijing Heyiyuan Biotech Co. Ltd. (Other); Shenzhen Microbiota Technology Co. Ltd. (Unknown)
Responsible Party: Principal Investigator, Fazheng Ren, Professor, China Agricultural University
Other Study IDs: CAUPCKD-01
Record Dates: First submitted 2016-12-28; First posted 2017-01-05 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Kidney Failure, Chronic
Keywords: Kidney Failure, Chronic; Uremic toxins; Gastrointestinal Microbiome; Metabolomics
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, serum, feces, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy subjects: Normal kidney function
  Interventions: Other: No interventions, questionnaire, collect specimen
- ESRD patients: Diagnosed as ESRD with hemodialysis
  Interventions: Other: No interventions, questionnaire, collect specimen

INTERVENTIONS:
Other: No interventions, questionnaire, collect specimen

SUMMARY:
The purpose of this study is to investigate the differences of gut Microbiome/Metabolite between ESRD patients and healthy subjects. Two hundred and twenty three hemodialysis patients and 70 healthy subjects are recruited, and a cross-sectional study is performed.

ELIGIBILITY:
For Healthy Subjects

Inclusion Criteria:

* Age over 18 years old
* Liver and kidney function is normal
* 18.5≤BMI≤29.9
* Agree to sign the informed consent form

Exclusion Criteria:

* Diagnosed as Metabolic syndrome
* Diagnosed as Cirrhosis
* Diagnosed as kidney disease
* Taking fermented food (live lactic acid bacteria drinks, cheese, yogurt, probiotic products, etc.) within 14 days before the study
* Taking antibiotics or antifungal drugs within 30 days before the study

For ESRD patients

Inclusion criteria:

* Age over 18 years old
* Patients who diagnosed as ESRD with hemodialysis
* Fixed hemodialysis cycle (average 3 times a week)
* Agree to sign the informed consent form

Exclusion criteria:

* Taking antibiotics or antifungal drugs within 30 days before the study
* Taking fermented food (live lactic acid bacteria drinks, cheese, yogurt, probiotic products, etc.) within 14 days before the study
* Reasercher are not sure whether the subjects are willing or able to complete the study
* Subject participated in other research projects within two months before the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two hundred and twenty three ESRD patients with hemodialysis are recruited from Department of Nephrology of 4 hospitals. Seventy healthy subjects are also recruited to compare the microbiome/metabolite differences between two groups.
Sampling Method: Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Microbiota-derived uremic toxin | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Fecal Microbiome | Through study completion, an average of 1 year
Fecal metabolites | Through study completion, an average of 1 year
Blood metabolites | Through study completion, an average of 1 year
Complete blood count | Through study completion, an average of 1 year
Blood biochemistry test | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Fazheng Ren, PhD, Principal Investigator — China Agricultural Universtiy
Locations (4):
- China (4):
  - Beijing Anzhen Hospital, Beijing
  - General Hospital of Chinese Armed Police Forces, Beijing
  - Peking University Aerospace Centre Hospital, Beijing
  - Peking University Shougang Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaziri ND, Wong J, Pahl M, Piceno YM, Yuan J, DeSantis TZ, Ni Z, Nguyen TH, Andersen GL. Chronic kidney disease alters intestinal microbial flora. Kidney Int. 2013 Feb;83(2):308-15. doi: 10.1038/ki.2012.345. Epub 2012 Sep 19. PMID 22992469
- [Background] Poesen R, Windey K, Neven E, Kuypers D, De Preter V, Augustijns P, D'Haese P, Evenepoel P, Verbeke K, Meijers B. The Influence of CKD on Colonic Microbial Metabolism. J Am Soc Nephrol. 2016 May;27(5):1389-99. doi: 10.1681/ASN.2015030279. Epub 2015 Sep 23. PMID 26400570
- [Background] Koppe L, Mafra D, Fouque D. Probiotics and chronic kidney disease. Kidney Int. 2015 Nov;88(5):958-66. doi: 10.1038/ki.2015.255. Epub 2015 Sep 16. PMID 26376131
- [Background] Anders HJ, Andersen K, Stecher B. The intestinal microbiota, a leaky gut, and abnormal immunity in kidney disease. Kidney Int. 2013 Jun;83(6):1010-6. doi: 10.1038/ki.2012.440. Epub 2013 Jan 16. PMID 23325079
- [Background] Ramezani A, Raj DS. The gut microbiome, kidney disease, and targeted interventions. J Am Soc Nephrol. 2014 Apr;25(4):657-70. doi: 10.1681/ASN.2013080905. Epub 2013 Nov 14. PMID 24231662
- [Background] Poesen R, Claes K, Evenepoel P, de Loor H, Augustijns P, Kuypers D, Meijers B. Microbiota-Derived Phenylacetylglutamine Associates with Overall Mortality and Cardiovascular Disease in Patients with CKD. J Am Soc Nephrol. 2016 Nov;27(11):3479-3487. doi: 10.1681/ASN.2015121302. Epub 2016 May 26. PMID 27230658
- [Background] Meyer TW, Hostetter TH. Uremia. N Engl J Med. 2007 Sep 27;357(13):1316-25. doi: 10.1056/NEJMra071313. No abstract available. PMID 17898101
- [Background] Aronov PA, Luo FJ, Plummer NS, Quan Z, Holmes S, Hostetter TH, Meyer TW. Colonic contribution to uremic solutes. J Am Soc Nephrol. 2011 Sep;22(9):1769-76. doi: 10.1681/ASN.2010121220. Epub 2011 Jul 22. PMID 21784895
- [Derived] Wang X, Yang S, Li S, Zhao L, Hao Y, Qin J, Zhang L, Zhang C, Bian W, Zuo L, Gao X, Zhu B, Lei XG, Gu Z, Cui W, Xu X, Li Z, Zhu B, Li Y, Chen S, Guo H, Zhang H, Sun J, Zhang M, Hui Y, Zhang X, Liu X, Sun B, Wang L, Qiu Q, Zhang Y, Li X, Liu W, Xue R, Wu H, Shao D, Li J, Zhou Y, Li S, Yang R, Pedersen OB, Yu Z, Ehrlich SD, Ren F. Aberrant gut microbiota alters host metabolome and impacts renal failure in humans and rodents. Gut. 2020 Dec;69(12):2131-2142. doi: 10.1136/gutjnl-2019-319766. Epub 2020 Apr 2. PMID 32241904